CLINICAL TRIAL: NCT04392102
Title: A Phase 2, Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of Niraparib in Patients With Advanced and Relapsed Ovarian Cancer After 3 or 4 Previous Chemotherapies
Brief Title: A Study of Niraparib in Patients With Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-2306-008
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZL-2306(Niraparib) (Experimental): The starting dose is 300mg or 200mg QD based on the subject's baseline body weight or baseline platelet count
  Interventions: Drug: ZL-2306(Niraparib）

INTERVENTIONS:
Drug: ZL-2306(Niraparib） — The starting dose is 300mg or 200mg QD based on the subject's baseline body weight or baseline platelet count
  Other Names: Zejula

SUMMARY:
This is a Phase 2, open-label, single arm study to evaluate the safety and efficacy of niraparib in ovarian cancer patients who have received three or four previous chemotherapy regimens. Niraparib is an orally active PARP inhibitor. Niraparib will be administered once daily continuously during a 28-day cycle. Health-related quality of life will be measured by Eastern Cooperative Oncology Group performance status (ECOG). Safety and tolerability will be assessed by clinical review of adverse events (AEs), physical examinations, electrocardiograms (ECGs), RECIST tumor assessments and safety laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must be female and at least 18 years of age
* 2. Patients must provide written informed consent
* 3. Patients must be gBRCA mutation or HRD positive
* 4. Patients must have histologically diagnosed high-grade (Grade 2 or 3)serous epithelial ovarian, fallopian tube, or primary peritoneal cancer with recurrent disease.
* 5. Patients Must have completed 3 or 4 previous chemotherapy regimens.
* 6. Patients must have measurable disease according to RECIST (v.1.1).
* 7. Patients must have an Eastern Cooperative Oncology Group(ECOG) performance status of 0 or1
* 8. Patients must have adequate organ function, defined as follows: a. Absolute neutrophil count≥1500/ul b. Platelets ≥150000/ul c. Hemoglobin≥10g/dL d. Serum creatinine≤1.5X upper limit of normal (ULN)or calculated creatinine clearance≥60ml/min using the Cockcroft-Gault equation e. Total bilirubin≤1.5X ULN OR direct bilirubin≤1X ULN f. Aspartate aminotransferase and alanine aminotransferase≤2.5X ULN unless liver metastases are present, in which case they must be ≤5X ULN
* 9. Patients must be either postmenopausal, free from menses for>12 months, surgically sterilized, or willing to use adequate contraception to prevent pregnancy or must agree to abstain from heterosexual activity throughout the study, starting with enrollment through 90 days after the last dose of study treatment
* 10. Patients must have formalin-fixed, paraffin-embedded tumor samples available form primary or recurrent cancer.
* 11. Patients must be able to take oral medications and capable of complying with treatment and follow up visit

Exclusion Criteria:

* 1. Patients who have received other investigational drugs within 4 weeks or 5X t1/2 before first dose of study treatment.
* 2. Patients have had palliative radiotherapy encompassing>20% of the bone marrow within 3 weeks of the first dose of study treatment.
* 3. Patients have any known, persistent(>4 weeks)，≥Grade 3 anemia, neutrophil count decrease or platelet count decrease during the last chemotherapy.
* 4. Patients have any known, persistent (>4 weeks), ≥ Grade 3 fatigue during the last chemotherapy.
* 5. Patients have received pelvic radiotherapy as treatment for primary or recurrent disease within 1 year of the first dose of study treatment.
* 6. Patients have symptomatic uncontrolled brain or leptomeningeal metastases. The patient have new or progressive signs or symptoms related to the CNS disease and not taking a stable dose of steroids or no steroids. A scan to confirm the absence of brain metastases is not required.
* 7. Patients have known hypersensitivity to the components of niraparib
* 8. Patient have had major surgery within 3 weeks of fist dose treatment and patient must have recovered form any effects of any major surgery
* 9. Patients have had diagnosis, detection, or treatment of invasive cancer other than ovarian cancer ≤2 years prior to enrollment(except basal or squamous cell carcinoma of the skin that has been definitively treated)
* 10. Patients are considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to: 1. uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction 2. uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome or any psychiatric disorder that prohibits obtaining informed consent 3. immune deficiency (not including splenectomy) 4. HIV infection or active hepatitis(i.e. hepatitis B with HBV-DNA>500IU/ml or hepatitis C with positive HCV-RNA).
* 11. Patients have received a transfusion (platelets or red blood cells) within 4 weeks of the first dose of study treatment.
* 12. Patients have known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* 13. Patients have current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study or interfere with patient's participation for the full duration of the study treatment or that makes it not in the best interest of the patient to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be female and at least 18 years of age
Enrollment: 15 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | Up to 3 years
  The ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) (version1.1).

SECONDARY OUTCOMES:
Duration of Response (DoR) | Up to 3 years
  DoR was defined as the time from first documentation of CR or PR until the time of first documentation of disease progression (PD) as assessed by the Investigator per RECIST (version1.1).
Disease Control Rate (DCR) | Up to 3 years
  Disease control rate was defined as the percentage of participants achieving CR, PR, or stable disease (SD) as assessed by the Investigator per RECIST (version1.1). The exact method was used to calculate 95% confidence interval.
Progression Free Survival (PFS) | Up to 3 years
  Progression-free survival was defined as the time from the date of first dose to the earlier date of assessment of progression or death by any cause in the absence of progression as assessed by the Investigator per RECIST (version 1.1).
Overall Survival (OS) | Up to 3 years
  Overall Survival was defined as the time from the date of the first dose to the date of death by any cause.
Number of Participants With Any Non-serious Adverse Event (Non-SAE) or Any SAE To evaluate the safety and tolerability of niraparib | Up to 3 years
  An adverse event is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly or birth defect or any other situation according to medical or scientific judgment was categorized as SAE.

CONTACTS AND LOCATIONS:
Overall Officials: Rutie Yin, Principal Investigator — West China Second University Hospital; Xiaohua Wu, Principal Investigator — Fudan University; Hong Zheng, Principal Investigator — Peking University Cancer Hospital & Institute; Ge Lou, Principal Investigator — Harbin Medical University; Lingying Wu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Hongmin Pan, Principal Investigator — Sir Run Shaw Hospital, school of medicine, Zhejiang University; Zhongqiu Lin, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University, Haerbin, Heilongjiang
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Second Iniversity Hospital, Chengdu, Sichuan
  - Sir Run Shaw Hospital, school of medicine, Zhejiang University, Guangzhou, Zhejiang